CLINICAL TRIAL: NCT02101463
Title: Surgeon-Modified Fenestrated/Branched Stent-Grafts for Treatment of Complex Aortic Aneurysms in High-Risk Patients
Brief Title: MOSTEGRA TRIAL:MO-(Dified) STE-(nt) GRA(-ft): Surgeon-modified Fenestrated-branched Stent-grafts
Acronym: MOSTEGRA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the organization and took the IDE/Study with him
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 997
Record Dates: First submitted 2014-03-25; First posted 2014-04-02 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Complex Aortic Aneurysms
Keywords: aortic; sm-FBSG; aneurysms; fenestrated; stent-grafts; Vascular; Endovascular
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgeon-modified fenestrated-branched stent-grafts (sm-FBSG) (Other)
  Interventions: Device: surgeon-modified fenestrated-branched stent-grafts (sm-FBSG)

INTERVENTIONS:
Device: surgeon-modified fenestrated-branched stent-grafts (sm-FBSG)

SUMMARY:
This trial evaluates surgeon-modified fenestrated-branched stent-grafts (sm-FBSG) for Abdominal Aortic Aneurysms (AAA) that are custom-made intra-operatively with no waiting period by a qualified vascular surgeon. In addition, it aims to examine the alternative sm-FBSG for patients with restricted access to centers performing clinical trials with commercially available devices and those patients with aortic emergencies.

DETAILED DESCRIPTION:
Complex aortic aneurysms are those involving the renal and visceral arteries, and open repair of these aneurysms requires more extensive dissection, aortic clamping above the renal or mesenteric arteries, and possible reconstruction of aortic branches. Recovery time tends to be longer, including more hospital days, than for endovascular repair, and there is a greater potential for complications. Many high-risk patients with aneurysms of the abdominal aorta (AAA), including thoracoabdominal aortic aneurysms (TAAA), and significant co-morbidities will be denied elective open surgery because of heightened risks associated with open repair of complex aneurysms, and therefore, the potential benefit of an endovascular option increases as well.

Endovascular aneurysm repair has been shown to be an effective alternative in treating uncomplicated infrarenal and thoracic aneurysms in both the elective and urgent setting, yet there is limited experience with this technology in complex conditions. Fenestrated grafts have been developed as a minimally invasive treatment for patients with complex aortic aneurysms who are unfit for traditional open surgery.

Surgeon-modified fenestrated-branch stent grafts (sm-FBSG) with branches for the visceral vessels are custom-made by a qualified vascular surgeon for patients with complex aortic conditions. It is expected that they will minimize surgical risks and promote quicker recovery, and they could represent a therapeutic option for high-risk patients unfit for open surgery.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

* Patients presenting for elective or urgent repair of a complex aortic aneurysm
* No other investigational agents or devices while on protocol
* Patient must be able and willing to comply with all follow-up exams
* Life expectancy of more than 1 year
* Patients with medical conditions that would make them unfit for open repair

Exclusion Criteria (abbreviated):

* Estimated life expectancy <1 year
* Contraindication to angiography
* Active infection
* Patients with ruptured or contained ruptured aortic aneurysm who are persistently hemodynamically unstable at the time of presentation
* Morbid Obesity with inability to visualize the aorta with available intraoperative imaging techniques

Anatomic exclusion criteria: iliac arteries and aorta must be able to accommodate endovascular devices and procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-08-28 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-12-08 (Actual)

PRIMARY OUTCOMES:
Determine the safety and effectiveness of sm-FBSG for the treatment of complex aortic aneurysms in patients at high-risk for open surgical repair. | 30 Days
  Major adverse events defined as:
  * All-cause death
  * Bowel ischemia
  * Myocardial infarction
  * Paraplegia
  * Renal failure
  * Respiratory failure
  * Stroke
  * Blood loss >=1,000cc
  The primary effectiveness endpoint is the proportion of treatment group subjects that achieve treatment success. Treatment success is a composite endpoint assessed at 12 months that includes successful delivery and deployment of the graft with branch vessel preservation (technical success) as well as freedom from Type 1 and 3 endoleaks, graft migration, and AAA enlargement or rupture.
  Technical success is defined as successful delivery and deployment of the physician modified endovascular graft with preservation of those branch vessels intended to be preserved. Includes freedom from the following at 12 months: Type I & III endoleak, stent graft migration, AAA enlargement, AAA rupture and conversion to open repair through 12 months.

SECONDARY OUTCOMES:
Evaluate postoperative all-cause morbidity after repair with sm-FBSG | >30 Days to 5 Years
  * Need for open surgical repair of the aortic aneurysm due to unsuccessful delivery or deployment of the stent graft for any reason
  * Internal bleeding or leaking of blood from the aneurysm subsequent to the index procedure
  * Organ dysfunction
Evaluate long-term survival and complications after repair of complex aortic aneurysms with sm-FBSG | >30 Days to 5 Years
  * Examination of Internal bleeding or leaking of blood from the aneurysm subsequent to the index procedure
  * Non-diagnostic intervention after the index procedure intended to correct or repair an endoleak, device migration, or other device defect.
  * Clinical evaluation and changes over time.
Successful device delivery and deployment with patency of all branches | 30 Days, 3 Months, 6 Months, and Years 1 to 5
  * Change in aneurysm sac diameter from the first post-procedural measurement; incidence of endoleak, device migration, or limb occlusion
  * Fenestrated stent graft patent luminal flow; absence of stent fracture or graft fatigue/failure
  * Renal and/or Mesenteric Artery and Stent Patency and Integrity
Procedural / In-Hospital Evaluations | 30 Days
  * Organ Perfusion and Function
  * Distal blood flow
  * Fluoroscopy time; contrast volume; estimated blood loss; % requiring transfusion; procedure time; ICU time; time to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Ricotta, II, MD, MS, FACS, Principal Investigator — Northside Hospital
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

REFERENCES:
- See also: Northside Vascular Website — http://www.nvs-ga.com/